CLINICAL TRIAL: NCT03155503
Title: A Single-center, Double-blind, Placebo-controlled, Randomized, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of SUVN-911 After Single Ascending Doses and Multiple Ascending Doses in Healthy Male Subjects
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of SUVN-911 in Healthy Subjects
Acronym: SUVN-911
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suven Life Sciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTP1S1911A4B2
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Depressive Disorder, Major
Keywords: SUVN-911; Depression; single dose; multiple dose; alpha4 beta2 receptor; first in human; safety; pharmacokinetics; tolerability
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: subjects randomized to drug or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single ascending dose (Active Comparator): Single dose of SUVN-911 or placebo in healthy male subjects
  Interventions: Drug: SUVN-911; Drug: Placebo
- Multiple ascending dose (Active Comparator): Multiple doses of SUVN-911 or placebo in healthy male subjects
  Interventions: Drug: SUVN-911; Drug: Placebo

INTERVENTIONS:
Drug: SUVN-911 — Oral Tablet
Drug: Placebo — Oral Tablet

SUMMARY:
This is a Phase 1, conventional, double-blind, placebo-controlled, single-center clinical study comprised of 2 segments (Segment 1 and Segment 2) in which single and multiple doses of SUVN-911 or placebo will be orally administered to healthy male subjects to evaluate the safety, tolerability, and pharmacokinetic profile.

DETAILED DESCRIPTION:
This is a single and multiple ascending dose study to assess the safety, tolerability and pharmacokinetics of SUVN-911 administered orally once a day to healthy male subjects. The study will be conducted under double-blind conditions.

The primary objectives are to evaluate the safety and tolerability of SUVN-911 following oral administration of single or multiple ascending doses and estimate the maximum tolerated dose of SUVN-911, if possible.

The secondary objectives are to evaluate the single and repeat dose plasma and urine pharmacokinetics of SUVN-911 following oral administration of single and multiple ascending doses in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged 18 to 45 years with a body mass index (BMI) between 18 and 30 kg/m2, (inclusive).

Exclusion Criteria:

* Standard exclusion criterion for Phase 1 clinical trial in healthy subjects:

  * History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate.
  * History or presence of gastro intestinal (GI), hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs as judged by Investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
ECG (Electrocardiogram) | Range of Day 1-17
  electrocardiogram outcomes
Vital signs | Range of Day 1-17
  blood pressure determination
C-SSRS (Columbia Suicidal Severity Rating Scale) | Range of Day 1-17
  Columbia Suicidal Severity Rating in multiple doses

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Day 1 and Day 14
  Plasma concentration
Maximum observed concentration (Cmax) | Day 1 and Day 14
  Maximum concentration observed
Time to reach maximum concentration (Tmax) | Day 1 and Day 14
  Determination of maximum time taken to reach the maximum concentration
Terminal half-life (t½) | Day 1 and Day 14
  Elimination rate

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lomeli, Principal Investigator — Quintiles, Inc.
Locations (1):
- QuintilesIMS Phase 1 Services, LLC, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nirogi R, Benade V, Goyal VK, Pandey SK, Mohammed AR, Shinde A, Dogiparti D, Ravula J, Jetta S, Palacharla VRC. Safety, Tolerability, and Pharmacokinetics of Ropanicant (SUVN-911), a Novel Alpha4 Beta2 Nicotinic Acetylcholine Receptor (alpha4beta2 nAChR) Antagonist, in Healthy Adult and Elderly Subjects. Clin Drug Investig. 2022 Sep;42(9):747-762. doi: 10.1007/s40261-022-01189-9. Epub 2022 Aug 13. PMID 35963959